CLINICAL TRIAL: NCT06941285
Title: Montreal Cognitive Assessment Index Following MRI Guided Focused Ultrasound
Brief Title: Montreal Cognitive Assessment Index Following MRI Guided Focused Ultrasound Thalamotomy
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ilana Schlesinger, Director Movement Disorders Institute, Rambam Health Care Campus
Other Study IDs: RMB0404-17
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
We assessed Montreal Cognitive Assessment scores before and after MRI guided focused ultrasound thalamotomy for tremor in order to identify if there are changes in cognitive function following treatment.

DETAILED DESCRIPTION:
All patients who underwent MRI guided focused ultrasound thalamotomy underwent cognitive assessment by Montreal Cognitive Assessment. We calculated the scores before and after treatment and compared the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent MRI guided focused ultrasound thalamotomy and suffered from Essential tremor.

Exclusion Criteria:

* Patients that did not undergo MRI guided focused ultrasound thalamotomy
* Patinets that did not suffer from Essential tremor.
* Patients that underwent MRI guided focused ultrasound for areas other then a thalamus
* Patients tat underwent bilateral thalamothomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent MRI guided focused ultrasound thalamotomy and suffered from Essential tremor.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | baselin, preprocedure, 6 months and 1 year
  Cognitive assessessment with higher score indicating better cognitive state

CONTACTS AND LOCATIONS:
Overall Officials: Inna Senderova, Study Director — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: Undecided